CLINICAL TRIAL: NCT03542916
Title: A Single-blind, Randomized, Single-dose, Crossover Study to Compare the Pharmacokinetics and Safety Following Administration of CJ-40001 and NESP® in Healthy Male Volunteers
Brief Title: Pharmacokinetics Study of CJ-40001 and NESP® After Single Dose Administration in Health Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CJ_EPO_101
Record Dates: First submitted 2015-01-26; First posted 2018-05-31 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2015-01

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CJ-40001 (Experimental): CJ-40001 60ug SC, IV injection
  Interventions: Drug: CJ-40001 60ug
- NESP (Active Comparator): NESP 60ug SC, IV injection
  Interventions: Drug: NESP 60ug

INTERVENTIONS:
Drug: CJ-40001 60ug — CJ-40001 60ug SC, IV injection
  Arms: CJ-40001
Drug: NESP 60ug — NESP 60ug SC, IV injection
  Arms: NESP

SUMMARY:
The purpose of this study is to compare the pharmacokinetics and safety after a single subcutaneous or intravenous administration of CJ-40001 and NESP® in healthy male volunteers.

DETAILED DESCRIPTION:
The purpose of this study is to compare the pharmacokinetics and safety after a single subcutaneous or intravenous administration of CJ-40001 and NESP in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 19 to 55 years at the screening
* Subject with BMI between 19 kg/m2 and 28 kg/m2 (inclusive)
* Subject who is able to participate in the whole study process
* Subject who provided written informed consent voluntarily after being fully informed of the study objectives, procedures and the investigational product

Exclusion Criteria:

* Subject who has a medical history of gastrointestinal, cardiovascular, respiratory, hepatobiliary, hematologic/oncologic, neuropsychologic, endocrinological, immunologic or renal disease that may be aggravated by the investigational product
* Subject with a systolic blood pressure of equal to or greater than 140 or less than 90 mmHg or with a diastolic blood pressure of equal to or greater than 90 or less than 60 mmHg
* Subject who has allergic disease that needs to be treated
* Subject with a history of drug allergies to any ingredient of the investigational product or marketed drug
* Subject with a blood hemoglobin value less than 13 g/dL or more than 17 g/dL
* Subject with a blood reticulocyte value more than the upper reference limit
* Subject with a blood vitamin B12 or ferritin or transferrin value less than the lower reference limit
* Subject with any non-negative results in blood serology (HBV, HCV, HIV, RPR) tests and in an examination of syphilis
* Subject who smokes more than 10 cigarettes per day
* Subject who consumes alcohol more than 140 g per week
* Subject with a history of drug abuse
* Subject who was administered with any investigational product, erythropoietin or iron supplement within 60 days prior to the screening
* Subject who donated whole blood within 60 days or blood components within 30 days prior to the screening
* Subject who took any herbal medicine within 30 days or any prescription drug within 14 days or over-the-counter drug considered to affect study within 10 days prior to the screening
* Subject who does not agree to use medically acceptable methods of contraception or who has plan to provide sperm during the study period
* Subject whom the investigator determined to have clinically significant findings in ECG
* Subject whose liver function is decreased with an AST, ALT or bilirubin value more than 1.5 times the upper reference limit
* Subject whose renal function is decreased with a GFR value calculated using MDRD equation less than the lower reference limit
* Subject whom the investigator determined to have clinically significant findings in clinical laboratory test
* Subject who is inappropriate as a subject of this study by the investigator's decision

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Assess Cmax of darbepoetin alfa in SC treatment group | SC treatment:Pre-dose and after dose up to 16 days
Assess Cmax of darbepoetin alfa in IV treatment group | IV treatment:Pre-dose and after dose 12 days
Assess AUClast of darbepoetin alfa in SC treatment group | SC treatment:Pre-dose and after dose up to 16 days
Assess AUClast of darbepoetin alfa in IV treatment group | IV treatment:Pre-dose and after dose 12 days

SECONDARY OUTCOMES:
Assess Temax of reticulocyte, hemoglobin, hematocrit, RBC in SC treatment group | SC treatment:Pre-dose and after dose up to 16 days
Assess Emax of reticulocyte, hemoglobin, hematocrit, RBC in SC treatment group | SC treatment:Pre-dose and after dose up to 16 days
Assess AUEClast of reticulocyte, hemoglobin, hematocrit, RBC in SC treatment group | SC treatment:Pre-dose and after dose up to 16 days
Assess Temax of reticulocyte, hemoglobin, hematocrit, RBC in IV treatment group | IV treatment:Pre-dose and after dose 12 days
Assess Emax of reticulocyte, hemoglobin, hematocrit, RBC in IV treatment group | IV treatment:Pre-dose and after dose 12 days
Assess AUEClast of reticulocyte, hemoglobin, hematocrit, RBC in IV treatment group | IV treatment:Pre-dose and after dose 12 days

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim S, Hong T, Ko JW, Huh W, Kim JR. Comparison of the Pharmacokinetic-Pharmacodynamic Relationships of Two Darbepoetin Alfa Formulations in Healthy Male Volunteers. BioDrugs. 2019 Feb;33(1):101-112. doi: 10.1007/s40259-018-0323-0. PMID 30506495